CLINICAL TRIAL: NCT03597074
Title: Diagnostic Value of Doppler Ultrasound for Early Prediction of Reversibility of Acute Kidney Injury in Septic ICU Patients
Brief Title: Doppler Ultrasound for Prediction of Reversibility of Acute Kidney Injury in Septic ICU Patients
Status: Completed | Type: Observational
Sponsor: Aristotle University Of Thessaloniki (Other)
Collaborators: George Papanicolaou Hospital (Other)
Responsible Party: Principal Investigator, Evangelos Kaimakamis, Principal Investigator, Aristotle University Of Thessaloniki
Other Study IDs: NT001
Record Dates: First submitted 2018-06-27; First posted 2018-07-24 (Actual); Last update posted 2018-07-24 (Actual); Status verified 2018-07

CONDITIONS: Acute Kidney Injury; Sepsis; Renal Resistive Index
Keywords: ICU; Renal Resistive Index; Acute Kidney Injury; Sepsis
MeSH Terms: conditions — Acute Kidney Injury; Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- 1: Patients without AKI progression Use of color Doppler Ultrasound derived Renal Resistive Index (RI) and semi-quantitative evaluation of intra-renal vascularization for early prognosis of AKI progression
  Interventions: Diagnostic Test: color Doppler Ultrasound derived RI and semi-quantitative evaluation of intra-renal vascularization
- 2: Patients with Transient AKI Use of color Doppler Ultrasound derived Renal Resistive Index (RI) and semi-quantitative evaluation of intra-renal vascularization for early prognosis of AKI progression
  Interventions: Diagnostic Test: color Doppler Ultrasound derived RI and semi-quantitative evaluation of intra-renal vascularization
- 3: Patients with Persistent AKI Use of color Doppler Ultrasound derived Renal Resistive Index (RI) and semi-quantitative evaluation of intra-renal vascularization for early prognosis of AKI progression
  Interventions: Diagnostic Test: color Doppler Ultrasound derived RI and semi-quantitative evaluation of intra-renal vascularization

INTERVENTIONS:
Diagnostic Test: color Doppler Ultrasound derived RI and semi-quantitative evaluation of intra-renal vascularization — Use of color Doppler Ultrasound derived Renal Resistive Index (RI) and semi-quantitative evaluation of intra-renal vascularization for early prognosis of AKI progression

SUMMARY:
Purpose: The aim of this study was to assess the ability of early discrimination between transient and persistent Acute Kidney Injury (AKI) using the color Doppler Ultrasound derived Renal Resistive Index (RI) and semi-quantitative evaluation of intra-renal vascularization in septic patients in an Intensive Care Unit (ICU).

Methods: Prospective observational cohort study with unselected, with 32 adult consecutive septic patients. Patients were divided into 3 groups: Group 1: patients without progression to AKI, Group 2: transient AKI, Group 3: persistent AKI.

DETAILED DESCRIPTION:
Purpose: The aim of this study was to assess the ability of early discrimination between transient and persistent AKI using the color Doppler Ultrasound derived Renal Resistive Index (RI) and semi-quantitative evaluation of intra-renal vascularization in septic patients in an Intensive Care Unit (ICU). Additionally, the investigators aimed to identify whether these indexes are early predictors of the prognosis of renal function in this group of patients. And compare the diagnostic accuracy of those and other renal indexes for the identification of AKI reversibility.

Methods: This was a prospective observational cohort study with unselected, consecutive septic patients included. Thirty-two adult septic patients hospitalized in a general ICU were studied. After the determination of sepsis, patients were divided into 3 groups: Group 1 included patients without progression to AKI, Group 2 included patients with transient AKI and Group 3 patients with persistent AKI.

ELIGIBILITY:
Inclusion Criteria:

* Septic patients in ICU
* Age 18 years or older

Exclusion Criteria:

* ICU stay less than 3 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects were included if they developed sepsis plus AKI during their hospitalization in the ICU, regardless of the underlying cause. The presence of Acute Kidney Injury was determined according to the KDIGO guidelines, i.e. at least stage 1 AKI. The categorization of AKI as transient or persistent was determined by the normalization of the kidney function after the administration of appropriate therapy and support in the ICU environment and after 3 days of hospitalization. All consecutive patients with sepsis were included, with the exception of those surviving less than three days, to determine whether they had AKI
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2017-03-02 (Actual); Primary Completion 2017-08-31 (Actual); Study Completion 2017-09-02 (Actual)

PRIMARY OUTCOMES:
RI as a prognostic factor for AKI persistence | 3 days
  without units (range 0 to 1)

SECONDARY OUTCOMES:
semi-quantitative US evaluation of renal vasculature | 3 days
  without units (score from 1 to 4)
FENa (Fractional Excretion of Sodium) | 3 days
  % percentage

CONTACTS AND LOCATIONS:
Overall Officials: Militsa Bitzani, MD, PhD, Study Director — 1st ICU, "G.Papanikolaou" General Hospital of Thessaloniki, Greece
Locations (1):
- 1st ICU, "G.Papanikolaou" General Hospital of Thessaloniki, Greece, Thessaloniki, Greece

IPD SHARING:
Plan to Share IPD: No
Data sheet can be shared with other researchers as soon as a publication of the results is achieved.

REFERENCES:
- [Background] Ninet S, Schnell D, Dewitte A, Zeni F, Meziani F, Darmon M. Doppler-based renal resistive index for prediction of renal dysfunction reversibility: A systematic review and meta-analysis. J Crit Care. 2015 Jun;30(3):629-35. doi: 10.1016/j.jcrc.2015.02.008. Epub 2015 Feb 24. PMID 25746587
- [Background] Schnell D, Deruddre S, Harrois A, Pottecher J, Cosson C, Adoui N, Benhamou D, Vicaut E, Azoulay E, Duranteau J. Renal resistive index better predicts the occurrence of acute kidney injury than cystatin C. Shock. 2012 Dec;38(6):592-7. doi: 10.1097/SHK.0b013e318271a39c. PMID 23042202

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-10-05): https://cdn.clinicaltrials.gov/large-docs/74/NCT03597074/Prot_SAP_000.pdf